CLINICAL TRIAL: NCT00928603
Title: Focal Therapy for Organ Confined Prostate Cancer: an Investigative Prospective Pilot Study
Brief Title: Investigative Study of the Role of Focal Therapy for Prostate Cancer Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Prof. Guazzoni Giorgio, Department of Urology, University "Vita Salute" San Raffaele Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-HSR-VT-001
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cryotherapy (Experimental): Focal Cryotherapy of localized tumor of prostate after spatial definition by in-house extended perineal core biopsy using a template biopsy strategy under local or general anesthesia
  Interventions: Procedure: Focal Cryoablation

INTERVENTIONS:
Procedure: Focal Cryoablation — Cryotherapy is administered via the perineum under ultrasound guidance by third-generation 17-gauge cryoprobes using gas and thermal couples. Under transrectal ultrasound guidance cryoprobes are placed approximately 1 cm apart and within 5 mm of the capsule on the side of tumor. The extent of freezing was limited to the area or lobe of the gland with histologically proved tumor.
  Other Names: Thermal ablative treatment

SUMMARY:
Surgery and irradiation for organ confined prostate cancer provide excellent long-term cancer control but they may be accompanied by a risk of side effects that decrease quality of life. Due to the stage migration of prostate cancer, the potential for patients to undergo unnecessary treatment and the risk of treatment related morbidity, has been increased.Alternative strategies that offer the possibility of delaying, obviating or minimizing the impact of treatment maintaining the same oncological long term results have been investigated. Despite pros and cons active surveillance has not gained popularity in men with low risk prostate cancer as only 7% of men with localized prostate cancer remain in active surveillance.

Traditionally solid tumors have been treated with radical surgery but selective, organ sparing therapies are now common for tumors of the breast, skin and kidney, resulting in equivalent rates of cancer control, lower morbidity rates and less disfigurement. With this in mind the potential role of focal ablative therapy for localized prostate cancer might be considered.

The researchers will investigate the feasibility and the efficacy in term of quality of life and oncologic results of focal therapy by a pilot not randomized prospective study in a patients with localized prostate cancer who meet low risk criteria based on clinical, biopsy and imaging data.

DETAILED DESCRIPTION:
Prostate cancer is a considerable health risk for men throughout the world. In the United States, prostate cancer has been the second or third leading cause of cancer death in men in each of the last 75 years. In the European Union, an estimated 68,000 men died of prostate cancer in 2004, making it the third most common cause of cancer related death While prostate cancer mortality in East Asian countries remains lower than that in Europe and the United States, it has been continuously and dramatically increasing in the last 40 years. With the introduction of PSA screening test and transrectal ultrasound guided prostate biopsy, the detection rate of prostate carcinoma has markedly improved. Surgery and irradiation each provide excellent long-term cancer control but they may be accompanied by a risk of side effects that decrease quality of life. Since some of prostate cancers grow slowly and, even if untreated, might never progress to symptomatic disease, patients and clinicians face the dilemma of if, when and how to treat localized prostate cancer. Due to the stage migration of prostate cancer, the potential for patients to undergo unnecessary treatment and the risk of treatment related morbidity, there has been, in the last years, an increased interest in alternative strategies that offer the possibility of delaying, obviating or minimizing the impact of treatment maintaining the same oncological long term results. One such strategy is active surveillance with selective delayed intervention. Active surveillance consists of appropriate selection of patients to safely avoid radical treatment and its attendant potential for morbidity, regular and rigorous monitoring of the cancer via physical examination, PSA, biopsies and imaging and initiation of treatment with curative intent at any clinical, pathological or radiographic evidence of disease progression. Despite pros and cons have recently addressed, active surveillance has not gained popularity in men with low risk prostate cancer (only around 7% of men with localized prostate cancer in the Cancer of the Prostate Strategic Urologic Research Endeavor national registry have elected to undergo active surveillance as the initial treatment options). Traditionally solid tumors have been treated with radical surgery but selective, organ sparing therapies are now common for tumors of the breast, skin and kidney, resulting in equivalent rates of cancer control, lower morbidity rates and less disfigurement. With this in mind the potential role of focal ablative therapy for localized prostate cancer might be considered. We investigate the feasibility and the efficacy in term of quality of life and oncologic results of focal therapy by a pilot not randomized prospective study in a patients with localized prostate cancer who meet low risk criteria based on clinical, biopsy and imaging data.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical

   * Clinical stage T1c or T2a
   * PSA less than 10 ng/ml
   * PSA velocity less than 2 ng/ml yearly in the year prior to diagnosis
2. Biopsy

   * Minimum of 12 cores
   * No Gleason grade 4 or 5
   * Maximum percentage of cancer in each core (20%)
   * Maximum length of cancer in each core ( 5 mm)
   * Maximum percentage of total cores with cancer (20%)
3. Imaging

   * Single lesion with a maximum size (12 mm)
   * Maximum length of capsular contact (10 mm)
   * No evidence of extraprostatic extension or seminal vesicle invasion

Exclusion Criteria:

1. Tumor in the transitional zone
2. Previous prostate surgery for benign pathology
3. Any rectal or perineal pathology hampering instrumentation and manipulation of the area
4. Benign or malignant rectal lesion
5. Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility, Safety, Tolerability (patient's complying with the follow-up), and Oncological efficacy | 5 years

SECONDARY OUTCOMES:
Changes in QoL instruments (IPSS/IIEF/FACT-P/MSHQ) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Guazzoni, MD, Study Director — University "Vita e Salute" San Raffaele Milano
Locations (1):
- Department of Urology University "Vita e Salute" HSR, Milan, Italy

REFERENCES:
- [Derived] Losa A, Gadda GM, Lazzeri M, Lughezzani G, Cardone G, Freschi M, Lista G, Larcher A, Nava LD, Guazzoni G. Complications and quality of life after template-assisted transperineal prostate biopsy in patients eligible for focal therapy. Urology. 2013 Jun;81(6):1291-6. doi: 10.1016/j.urology.2012.11.078. Epub 2013 Mar 19. PMID 23522299